CLINICAL TRIAL: NCT06882161
Title: Clinical and Radiographic Evaluation of The Effect of Acetal Resin Versus PEEK on Supporting Structure of Abutment Teeth in Mandibular Kennedy Class I Partial Dentures Manufactured by CAD-CAM Technology
Brief Title: Clinical and Radiographic Evaluation of The Effect of Acetal Resin Versus PEEK on Supporting Structure of Abutment Teeth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Yasmin Seif Eldeen Zidan, Yasmin S. Zidan, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: P-PD-14-14
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — acetalic resin, Acetal-Dental; polyetheretherketone

STUDY DESIGN:
Intervention Model Description: This study was a parallel, two-group, double-blinded, randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: (patients and assessors)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetal resin partial dentures (Active Comparator): ten patients received acetal resin partial dentures designed and fabricated using CAD/CAM technology
  Interventions: Biological: Acetal resin
- PEEK partial dentures (Active Comparator): ten patients received polyether ether ketone (PEEK) partial dentures designed and fabricated using CAD/CAM technology.
  Interventions: Biological: Acetal resin

INTERVENTIONS:
Biological: Acetal resin — Effect of acetal resin versus Polyether ether ketone (PEEK) partial dentures on abutment teeth supporting structures in Kennedy class I mandibular partial denture cases
  Other Names: PEEK

SUMMARY:
This study was conducted to evaluate and compare the effect of acetal resin versus Polyether ether ketone (PEEK) partial dentures on abutment teeth supporting structures in Kennedy class I mandibular partial denture cases. Clinical assessments were conducted by assessing the pocket depth (PD), plaque index (PI), and gingival index (GI). Cone beam computed tomography (CBCT) was used to assess abutment alveolar bone height change.

DETAILED DESCRIPTION:
This study was a parallel, two-group, double-blinded, randomized clinical trial. The proposal and consents were approved by the Research Ethics Committee. (REC) approval (P-PD-14-14). The Helsinki Declaration's guiding principles were followed when conducting the study. The Comprehensive Standards of Reporting Trials Statement (CONSORT) checklist's structure is followed in the study's presentation. The study was carried out at the Outpatient Clinic of the Removable Prosthodontic Department within the Faculty of Dental Medicine for Girls at Al-Azhar University.

In this study, fifty patients were initially evaluated. After conducting clinical and radiographic assessments, twenty patients who satisfied the inclusion criteria were selected in accordance with the sample size calculation. Each patient received an explanation of every procedure, and informed consent was obtained. These twenty individuals were subsequently divided randomly into two distinct groups (ten in each):

Group I: Ten patients received polyoxymethylene (acetal resin) partial dentures designed and fabricated using CAD/CAM technology. Group II: Ten patients received polyether ether ketone (PEEK) partial dentures designed and fabricated using CAD/CAM technology.

All patients were evaluated clinically and radiographically. Clinical assessments were conducted by assessing the pocket depth (PD), plaque index (PI), and gingival index (GI) at denture insertion, three months later and six months later. Cone beam computed tomography (CBCT) was used to assess abutment alveolar bone height change at the time of denture placement, after three months, and after six months.

ELIGIBILITY:
Inclusion Criteria:

* Every subject should be free of any systemic diseases that might influence the results of the research.
* Patient's residual ridges should be covered with healthy mucosa.
* Their salivary flow and viscosity for all within normal limits.
* The patients are cooperative and ready to be called back as necessary.
* had a Class I Angle's ridge relation

Exclusion Criteria:

* Alcoholic or smokers' patients.
* Patients with xerostomia or excessive salivation.
* Patients with parafunctional habits.
* Patients with ulcerated or inflamed mucosa.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Pocket Depth | 6 months
  assessing the pocket depth (PD) of abutment teeth

SECONDARY OUTCOMES:
Plaque index | 6 months
  assessing the plaque index (PI) of abutment teeth
Gingival index | 6 months
  assessing the gingival index (GI) of abutment teeth
Abutment alveolar bone height change. | 6 months
  assessing the Abutment alveolar bone height of abutment teeth

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin S Zidan, PhD, Principal Investigator — Lecturer at faculty of dental medicine for girls , Al-Azhar University
Locations (1):
- Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No